CLINICAL TRIAL: NCT04615039
Title: Post Market Clinical Follow-Up Study for MicroPort PROFEMUR® Preserve Classic Femoral Stem
Status: Withdrawn | Type: Observational
Why Stopped: Site selection process has been revisited
Sponsor: MicroPort Orthopedics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19H001C
Record Dates: First submitted 2020-10-22; First posted 2020-11-04 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Joint Diseases
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: PROFEMUR® Preserve Classic Femoral Stem — Single study group of subjects, either newly or previously implanted with the PROFEMUR® Preserve Classic Femoral Stem combined with any type of polyethylene and ceramic acetabular shells, acetabular liners and femoral heads.

SUMMARY:
Sponsor is conducting this post market clinical study to evaluate the safety and effectiveness of its PROFEMUR® Preserve Classic Femoral Stem. This type of study is required by regulatory authorities for all devices that have been approved in Europe (EU) to evaluate the medium and long-term clinical evidence. This study has been designed in accordance with MEDDEV2.12/2 (European Medical Device Vigilance System) rev2 and ISO (International Organization of Standardization) 14155:2011 guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Has previously undergone or currently has been determined to undergo a primary THA with the study component MPO PROFEMUR® Preserve Classic Stem combined with any type of polyethylene or ceramic acetabular shells, acetabular liners and femoral heads.
2. Has previously undergone or currently has been determined to undergo a primary THA for any of the following:

   * non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, ankylosis, protrusio acetabuli, and painful hip dysplasia;
   * inflammatory degenerative joint disease such as rheumatoid arthritis;
   * correction of functional deformity
3. Willing and able to complete required study visits and assessments through the 10 year postoperative follow-up visit.
4. Previously implanted subjects must be enrolled within 3 years (+ 6 months) of their primary THA implantation.

Exclusion Criteria:

1. Skeletally immature (less than 21 years of age) at time of implantation
2. Has or had an overt infection at the time of implantation
3. Has or had a distant foci of infections (which may cause hematogenous spread to the implant site) at the time of implantation
4. Has or had a rapid disease progression as manifested by joint destruction or bone absorption apparent on roentgenogram at the time of implantation
5. Has or had inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable
6. Has or had neuropathic joints
7. Has or had hepatitis or HIV infection
8. Has or had a neurological or musculoskeletal disease that may adversely affect gait or weight-bearing
9. Has or had a revision procedure(s) where other treatments or devices have failed; and treatment of fractures that are unmanageable using other techniques
10. Currently enrolled in another clinical investigation which could affect the endpoints of this protocol
11. Has or had documented substance abuse issues
12. Has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
13. Currently incarcerated or has impending incarceration
14. Has a medical condition, as judged by the Investigator, that would interfere with the subject's ability to comply with the requirements of the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with either newly or previously implanted with the PROFEMUR® Preserve Classic Femoral Stem combined with any type of polyethylene and ceramic acetabular shells, acetabular liners and femoral heads.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Component Survivorship | 10 years post-operative
  To estimate component survivorship of the PROFEMUR® Preserve Classic Femoral Stem at 1, 3, 5, 7, 10 years.

SECONDARY OUTCOMES:
HOOS Functional Scores | 10 years post-operative
  Complete characterization (mean, minimum, maximum, standard deviation) of functional scores as assessed by the Hip Disability and Osteoarthritis Outcome Score (HOOS), which ranges from 0 to 100 with a score of 0 indicating worst hip symptoms and 100 indicating no hip symptoms.
EQ-5D-5L Functional Scores | 10 years post-operative
  Complete characterization (mean, minimum, maximum, standard deviation) of functional scores as assessed by EQ-5D-5L. This functional score data will be summarized over 5 domains, namely, mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain has 5 levels: no problems, slight problem, moderate problem, severe problem, inability to perform the activity. With no problems being the best outcome and inability to perform the activity being worst outcome.
Subject Satisfaction as assessed by Forgotten Joint Score | 10 years post-operative
  To determine proportion of subjects being satisfied and level of their satisfaction as assessed by the Forgotten Joint Score (FJS). The study will be reporting forgotten joint score measures for the assessment of joint-specific patient reported outcomes. The questions focus on the patients' awareness of the implanted joint in everyday life or any unintended perception of a joint.
Subject Satisfaction as assessed by Satisfaction Survey | 10 years post-operative
  To determine proportion of subjects being satisfied and level of their satisfaction as assessed by the Satisfaction Survey, consisting of questions asked about how satisfied the patient is with the new implant.
Radiolucencies | 10 years post-operative
  To assess the presence of radiolucencies surrounding implanted components
To assess subject safety | 10 years post-operative
  To assess safety of the PROFEMUR® Preserve Classic Femoral Stem through device-related adverse event findings and/or adverse device effects during follow-up visits.
To assess device tolerability within subject | 10 years post-operative
  To assess tolerability of the PROFEMUR® Preserve Classic Femoral Stem through device-related adverse event findings and/or adverse device effects during follow-up visits.

IPD SHARING:
Plan to Share IPD: No